CLINICAL TRIAL: NCT02260726
Title: Diagnosing Deformities of the Hip Associated With Arthritis: MRI vs Ultrasound
Brief Title: Evaluation of Ultrasound for Detecting Hip Impingement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding available
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20140318-01H
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Femoroacetabular Impingement
Keywords: femoroacetabular impingement; morphometry; dynamic; magnetic resonance imaging; ultrasound; screening; diagnosis
MeSH Terms: conditions — Femoracetabular Impingement; Disease | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical group (Experimental): Subjects already scheduled to undergo surgical correction of a symptomatic cam-type hip impingement deformity. Subjects will undergo magnetic resonance imaging (MRI) and ultrasound investigation prior to surgery.
  Interventions: Procedure: Magnetic resonance imaging; Procedure: Ultrasound
- Control (Other): Asymptomatic subjects with normal hip morphometry, as determined by MRI. Subjects will undergo magnetic resonance imaging (MRI) and ultrasound imaging.
  Interventions: Procedure: Magnetic resonance imaging; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Magnetic resonance imaging
Procedure: Ultrasound

SUMMARY:
Patients are being asked to participate in this study because a previous research MRI of their hips showed that the shape of the head of their thigh bone may indicate FAI of the hip. We have already collected cartilage imaging data and data on how the hip joint moves on people with painful/symptomatic FAI and people with normal hip function. We would now like to compare the motion of the hip joint to those with painful FAI using ultrasound.

DETAILED DESCRIPTION:
Hip impingement is thought to be a leading cause of hip osteoarthritis, and occurs due to deformities in the hip joint. However some individuals have these deformities but do not exhibit symptoms. Using the standard magnetic resonance imaging and clinical tests it is not clear which deformities will cause degeneration, requiring surgical intervention. We propose to evaluate the deformity and impingement between the femur and acetabulum using dynamic ultrasound imaging. Ultrasound does not involve radiation and can acquire video of the hip joint and is thus suitable for such diagnostic purposes. In this pilot study we will evaluate the feasibility of ultrasound in diagnosing hip impingement.

ELIGIBILITY:
Inclusion Criteria:

Surgical group:

* Hip pain longer than 6 months referred to the groin/lateral aspect of the hip
* Positive Impingement Sign

Plain radiographs:

* Absence of arthritis (Tonnis Grade 0 or 1)
* Absence of dysplasia (center edge >25 degrees) on anterior-posterior radiograph
* α-angle greater than 60 degrees on MRI.

Exclusion Criteria:

* Patients who don't meet inclusion criteria
* Control group: subjects with hip pain or with alpha angle > 50 degrees on MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10 (Estimated); Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Ultrasound grade | Upon enrollment
  Ultrasound grade evaluated on a four point scale following ultrasound imaging session

SECONDARY OUTCOMES:
Ultrasound parameters | Upon enrollment
  Morphometry of hip measured in ultrasound images: alpha angle, clearance angle
MRI parameters | Upon enrollment
  Standard MRI measures of impingement from images. Used as gold standard for comparative purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — University of Ottawa / The Ottawa Hospital